CLINICAL TRIAL: NCT05521165
Title: Effect of Gluteus Medius Strengthening on Pain, Function, and Muscle Macromorphology in Nonspecific Chronic Low Back Pain
Brief Title: Gluteus Medius Strengthening n Non Specific Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadil Mohamed Onsy Mohamed Salama, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gluteus Medius in back pain
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Gluteus Medius, Ultrasonography, NSCLBP
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): The patients in group (A) (n=29) will receive an American physical therapy association (APTA) guided program consisting of stretching exercises for global trunk, back muscles, and hamstring muscles, strengthening exercises for abdominal and back muscles, and stabilizing exercises for trunk and pelvic muscles.
  Interventions: Other: therapeutic exercises
- group B (Experimental): The patients in group (B) (n=29) will receive treatment as in group (A) in addition to selected G Med strengthening exercises.
  Interventions: Other: therapeutic exercises

INTERVENTIONS:
Other: therapeutic exercises — strengthening exercises for gluteus medius and APTA guided program for NSCLBP

SUMMARY:
To study the effect of adding selected G Med muscle strengthening exercises to the APTA-guided program on pain, disability level, and G Med macromorphology in patients with NSCLBP.

DETAILED DESCRIPTION:
Low back pain (LBP) is a significant global health problem. It occurs in all age groups from children to the elderly. Costs associated with health care and work disability attributed to LBP vary between countries and are influenced by social and health care approaches.

In almost all people with LBP, it is not possible to identify a specific cause. Only a small proportion of people have a well-understood pathological reason e.g., a vertebral fracture, malignancy, or infection. On the other hand, non-specific chronic low back pain (NSCLBP) accounts for about 85% of LBP patients treated in primary care, and the vast majority of patients with LBP seen by physical therapists are classified under this designation.

A recently published systematic review examined the impairment of lower extremity muscle strength in LBP disorders. The researchers reported a significant reduction in hip abductor, extensor, and knee extensor strength in patients with LBP compared to their healthy controls.

Researchers examined the strength of gluteus medius (G Med) muscle function in patients with LBP compared to non-LBP controls. The study reported that G Med muscle strength was decreased and several trigger points were developed but there were unclear results on fatigability, activity level, and macromorphology compared to healthy individuals.

It was evident, however, that the slight increase in muscle thickness of certain local and global muscles during contraction in the NSCLBP group compared to a healthy group when examined by ultrasonography could be an indicator that the strengthening of the multifidus, the transversus abdominis, and the G Med prevents the occurrence of LBP.

Exercise therapy is one of the inexpensive tools addressing pain relief and disability management in patients with subacute, chronic low back pain (CLBP) compared to usual care, according to the recently published systematic review.

Various types of exercise interventions should be used by physical therapists in the management of CLBP, as recommended by the American Physical Therapy Association (APTA) guidelines for clinical practice.

In a study by Mendis & Hides (2016), they demonstrated lumbar-pelvic muscle imbalance in LBP and improvement in sartorius and G Med muscle size when motor training interventions were applied in non-weight-bearing and weight-bearing positions during treatment of LBP.

A recent study evaluated the effectiveness of adding specific hip strengthening exercises to a conventional rehabilitation program in the management of LBP patients. The results of the systematic review revealed that hip strengthening exercises could reduce pain and disability in these patients.

At the same time, there is still a knowledge gap regarding the effect of G Med strengthening exercise specifically on pain and disability levels in patients with NSCLBP and muscle macromorphology (thickness), as recommended in several recent systematic reviews.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged between 20-45yrs 2. Patients with NSCLBP (pain > 3 months). 3. NSCLBP must have been present for at least the previous 12 weeks. 4. Patients with unilateral or bilateral symptoms that are worse on one side than the other, are referred by an orthopedist.

Exclusion Criteria:

* 1. 'Red Flag' symptoms include, a history of major trauma, persistent night pain, bladder or bowel dysfunction, and/or lower extremity neurological deficit.

  2. History of previous back surgery. 3. History of the previous pelvis or hip surgeries. 4. Recent or old fractures in lower limbs. 5. Cognitive impairment and inability to understand the scale. 6. Systemic inflammatory diseases e.g., rheumatoid arthritis and ankylosing spondylitis.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
back Pain intensity level | 6 weeks
  The Numerical Pain Rating Scale (NPRS) for pain is a one-dimensional measure of pain intensity.
disability level of low back pain patients | 6 weeks
  Back pain related disability is estimated using the cross-culturally adapted Arabic version of Oswestry disability index (ODI-AR).
G Med macromorphology | 6 weeks
  measuring gluteus medius thickness by ultrasonography

REFERENCES:
- [Background] Abe T, Loenneke JP, Thiebaud RS. Morphological and functional relationships with ultrasound measured muscle thickness of the lower extremity: a brief review. Ultrasound. 2015 Aug;23(3):166-73. doi: 10.1177/1742271X15587599. Epub 2015 May 29. PMID 27433253
- [Background] Aboufazeli M, Akbari M, Jamshidi AA, Jafarpisheh MS. Comparison of Selective Local and Global Muscle Thicknesses in Females with and without Chronic Low Back Pain. Ortop Traumatol Rehabil. 2018 Jun 27;20(3):197-204. doi: 10.5604/01.3001.0012.1473. PMID 30152768
- [Background] Algarni AS, Ghorbel S, Jones JG, Guermazi M. Validation of an Arabic version of the Oswestry index in Saudi Arabia. Ann Phys Rehabil Med. 2014 Dec;57(9-10):653-63. doi: 10.1016/j.rehab.2014.06.006. Epub 2014 Aug 4. PMID 25262247
- [Background] Amabile AH, Bolte JH, Richter SD. Atrophy of gluteus maximus among women with a history of chronic low back pain. PLoS One. 2017 Jul 17;12(7):e0177008. doi: 10.1371/journal.pone.0177008. eCollection 2017. PMID 28715424
- [Background] Ayotte NW, Stetts DM, Keenan G, Greenway EH. Electromyographical analysis of selected lower extremity muscles during 5 unilateral weight-bearing exercises. J Orthop Sports Phys Ther. 2007 Feb;37(2):48-55. doi: 10.2519/jospt.2007.2354. PMID 17366959
- [Background] Bernet BA, Peskura ET, Meyer ST, Bauch PC, Donaldson MB. The effects of hip-targeted physical therapy interventions on low back pain: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2019 Feb;39:91-100. doi: 10.1016/j.msksp.2018.11.016. Epub 2018 Dec 1. PMID 30553988
- [Background] Cooper NA, Scavo KM, Strickland KJ, Tipayamongkol N, Nicholson JD, Bewyer DC, Sluka KA. Prevalence of gluteus medius weakness in people with chronic low back pain compared to healthy controls. Eur Spine J. 2016 Apr;25(4):1258-65. doi: 10.1007/s00586-015-4027-6. Epub 2015 May 26. PMID 26006705
- [Background] de Jesus FLA, Fukuda TY, Souza C, Guimaraes J, Aquino L, Carvalho G, Powers C, Gomes-Neto M. Addition of specific hip strengthening exercises to conventional rehabilitation therapy for low back pain: a systematic review and meta-analysis. Clin Rehabil. 2020 Nov;34(11):1368-1377. doi: 10.1177/0269215520941914. Epub 2020 Jul 21. PMID 32691625